CLINICAL TRIAL: NCT05932745
Title: Examining Appeal and Addiction Potential of Novel E-cigarette Constituents Among Adults
Brief Title: Effects of Novel E-cigarette Constituents on Adults TCORS 3.0
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2000035551_b; 2U54DA036151-11 (NIH)
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Nicotine Use Disorder
Keywords: Menthol, cooling components, cigarette, e-cigarette, vaping
MeSH Terms: conditions — Tobacco Use Disorder; Vaping | interventions — Menthol

STUDY DESIGN:
Intervention Model Description: All participants receive all 18 study conditions.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be given a nicotine containing e-cigarette that could have various levels of cooling flavoring. Participants will not be told the nicotine concentration of the product or the type or concentration of the added coolant or what order it is presented in. Investigator and research assistant (i.e. care provider) will know the doses of nicotine and coolant, but will not know what order coolants are presented to participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (18):
- Non-menthol, nicotine 59mg/ml (1) (Experimental): Flavor without menthol with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (No WS-3) for non-menthol (1)
- Low (0.1%) menthol, nicotine 59mg/ml (1) (Experimental): Flavor with low menthol concentration with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (No WS-3) for low (0.1%) menthol (1)
- High (2.0%) menthol, nicotine 59mg/ml (1) (Experimental): Flavor with high menthol concentration with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (No WS-3) for high (2.0%) menthol (1)
- Non-menthol, nicotine 59mg/ml (2) (Experimental): Flavor without menthol with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (Low [0.1%] WS-3) for non-menthol (2)
- Low (0.1%) menthol, nicotine 59mg/ml (2) (Experimental): Flavor with low menthol concentration with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (Low [0.1%] WS-3) for low (0.1%) menthol (2)
- High (2.0%) menthol, nicotine 59mg/ml (2) (Experimental): Flavor with high menthol concentration with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (Low [0.1%] WS-3) for high (2.0%) menthol (2)
- Non-menthol, nicotine 59mg/ml (3) (Experimental): Flavor without menthol with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (High [2.0%] WS-3) for non-menthol (3)
- Low (0.1%) menthol, nicotine 59mg/ml (3) (Experimental): Flavor with low menthol concentration with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (High [2.0%] WS-3) for low (0.1%) menthol (3)
- High (2.0%) menthol, nicotine 59mg/ml (3) (Experimental): Flavor with high menthol concentration with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (High [2.0%] WS-3) for high (2.0%) menthol (3)
- Non-menthol, nicotine 59mg/ml (4) (Experimental): Flavor without menthol with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (Low [0.1%] WS-23) for non-menthol (4)
- Low (0.1%) menthol, nicotine 59mg/ml (4) (Experimental): Flavor low menthol concentration with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (Low [0.1%] WS-23) for low (0.1%) menthol (4)
- High (2.0%) menthol, nicotine 59mg/ml (4) (Experimental): Flavor high menthol concentration with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (Low [0.1%] WS-23) for high (2.0%) menthol (4)
- Non-menthol, nicotine 59mg/ml (5) (Experimental): Flavor without menthol with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (High [2.0%] WS-23) for non-menthol (5)
- Low (0.1%) menthol, nicotine 59mg/ml (5) (Experimental): Flavor low menthol concentration with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (High [2.0%] WS-23) for low (0.1%) menthol (5)
- High (2.0%) menthol, nicotine 59mg/ml (5) (Experimental): Flavor high menthol concentration with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (High [2.0%] WS-23) for high (2.0%) menthol (5)
- Non-menthol, nicotine 59mg/ml (6) (Experimental): Flavor without menthol with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (4% WS-23) for non-menthol (6)
- Low (0.1%) menthol, nicotine 59mg/ml (6) (Experimental): Flavor low menthol concentration with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (4% WS-23) for low (0.1%) menthol (6)
- High (2.0%) menthol, nicotine 59mg/ml (6) (Experimental): Flavor high menthol concentration with 59mg/ml nicotine
  Interventions: Other: E-liquid coolant (4% WS-23) for high (2.0%) menthol (6)

INTERVENTIONS:
Other: E-liquid coolant (No WS-3) for non-menthol (1) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants without WS-3.
  Other Names: Flavor type
  Arms: Non-menthol, nicotine 59mg/ml (1)
Other: E-liquid coolant (No WS-3) for low (0.1%) menthol (1) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants without WS-3.
  Other Names: Flavor type
  Arms: Low (0.1%) menthol, nicotine 59mg/ml (1)
Other: E-liquid coolant (No WS-3) for high (2.0%) menthol (1) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants without WS-3.
  Other Names: Flavor type
  Arms: High (2.0%) menthol, nicotine 59mg/ml (1)
Other: E-liquid coolant (Low [0.1%] WS-3) for non-menthol (2) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with low WS-3 concentration.
  Other Names: Flavor type
  Arms: Non-menthol, nicotine 59mg/ml (2)
Other: E-liquid coolant (Low [0.1%] WS-3) for low (0.1%) menthol (2) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with low WS-3 concentration.
  Other Names: Flavor type
  Arms: Low (0.1%) menthol, nicotine 59mg/ml (2)
Other: E-liquid coolant (Low [0.1%] WS-3) for high (2.0%) menthol (2) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with low WS-3 concentration.
  Other Names: Flavor type
  Arms: High (2.0%) menthol, nicotine 59mg/ml (2)
Other: E-liquid coolant (High [2.0%] WS-3) for non-menthol (3) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with high WS-3 concentration.
  Other Names: Flavor type
  Arms: Non-menthol, nicotine 59mg/ml (3)
Other: E-liquid coolant (High [2.0%] WS-3) for low (0.1%) menthol (3) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with high WS-3 concentration.
  Other Names: Flavor type
  Arms: Low (0.1%) menthol, nicotine 59mg/ml (3)
Other: E-liquid coolant (High [2.0%] WS-3) for high (2.0%) menthol (3) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with high WS-3 concentration.
  Other Names: Flavor type
  Arms: High (2.0%) menthol, nicotine 59mg/ml (3)
Other: E-liquid coolant (Low [0.1%] WS-23) for non-menthol (4) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with low WS-23 concentration.
  Other Names: Flavor type
  Arms: Non-menthol, nicotine 59mg/ml (4)
Other: E-liquid coolant (Low [0.1%] WS-23) for low (0.1%) menthol (4) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with low WS-23 concentration.
  Other Names: Flavor type
  Arms: Low (0.1%) menthol, nicotine 59mg/ml (4)
Other: E-liquid coolant (Low [0.1%] WS-23) for high (2.0%) menthol (4) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with low WS-23 concentration.
  Other Names: Flavor type
  Arms: High (2.0%) menthol, nicotine 59mg/ml (4)
Other: E-liquid coolant (High [2.0%] WS-23) for non-menthol (5) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with high WS-23 concentration.
  Other Names: Flavor type
  Arms: Non-menthol, nicotine 59mg/ml (5)
Other: E-liquid coolant (High [2.0%] WS-23) for low (0.1%) menthol (5) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with high WS-23 concentration.
  Other Names: Flavor type
  Arms: Low (0.1%) menthol, nicotine 59mg/ml (5)
Other: E-liquid coolant (High [2.0%] WS-23) for high (2.0%) menthol (5) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with high WS-23 concentration.
  Other Names: Flavor type
  Arms: High (2.0%) menthol, nicotine 59mg/ml (5)
Other: E-liquid coolant (4% WS-23) for non-menthol (6) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with 4% WS-23 concentration.
  Arms: Non-menthol, nicotine 59mg/ml (6)
Other: E-liquid coolant (4% WS-23) for low (0.1%) menthol (6) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with 4% WS-23 concentration.
  Arms: Low (0.1%) menthol, nicotine 59mg/ml (6)
Other: E-liquid coolant (4% WS-23) for high (2.0%) menthol (6) — Adult users of e-cigarette will be exposed to distinct e-liquid coolants with 4% WS-23 concentration.
  Arms: High (2.0%) menthol, nicotine 59mg/ml (6)

SUMMARY:
This study is an examination of the influence of cooling components of WS-3, WS-23, and menthol on the appeal and addiction potential of nicotine-containing e-liquids among adults.

DETAILED DESCRIPTION:
The investigators will examine the influence of cooling components of WS-3, WS-23 (synthetic coolants) and menthol on the appeal and addiction potential of nicotine-containing e-liquids among adults. Participants will rate the flavor intensity, coolness, sweetness, and irritation/harshness, bitterness experienced using validated rating scales. 66 adult participants (18+ years of age) who are current e-cigarette users will participate in 3 laboratory sessions. Participants will be randomized to receive one of the 3 menthol conditions (no-menthol, low menthol, high menthol) in Lab 1 and will receive the alternative conditions in randomized order in Lab 2 and Lab 3. During each lab session the menthol condition will be paired with three WS-3 concentrations: no WS-3, low (0.1%) WS-3, or high (2.0%) WS-3 and three WS-23 concentrations: low (0.1%) WS-23, high (2.0%) WS-23, or 4% WS-23 in randomized order. All e-cigarettes will contain nicotine salt at a nicotine concentration of ~59mg/ml and all participants will be exposed to eighteen conditions across 3 lab sessions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to read and write
* Some current e-cigarette use
* Urine cotinine ≥200ng/ml
* Willing to abstain from tobacco/nicotine use 2 hours prior to sessions

Exclusion Criteria:

* Current use of non-prescription substances besides nicotine, marijuana, alcohol
* Any significant current medical or psychiatric condition
* Known hypersensitivity to propylene glycol
* Pregnant or lactating females
* Uncontrolled asthma
* Nut/e-liquid flavorant allergy
* Current marijuana (tetrahydrocannabinol) vaping + E-cigarette or vaping use Associated Lung Injury (EVALI) symptoms
* Dislike of menthol flavor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Liking: Score change in liking/wanting of each e-cigarette condition (5 conditions in total) | Following administration of e-cigarette condition 1 (at 10 minutes), following administration of e-cigarette condition 2 (at 40 minutes)...following administration of e-cigarette condition 6 (at 160 minutes)
  The Labeled Hedonic Scale will be used to ask about liking and wanting of the e-cigarette (one item Visual Analog Scale with ratings ranging from "most disliked sensation imaginable" to "most liked sensation imaginable" with higher values indicating greater liking).
Reinforcing Efficacy: Score change in drug effects of each e-cigarette condition (5 conditions in total) | Following administration of e-cigarette condition 1 (at 10 minutes), following administration of e-cigarette condition 2 (at 40 minutes)...following administration of e-cigarette condition 6 (at 160 minutes)
  Difference between e-cigarette effects for each e-cigarette condition as measured by the computerized version of the Drug Effects Questionnaire (DEQ). Participants will self-report their responses using a computer mouse to indicate where on the scale response falls. A modified version of the Drug Effects Questionnaire (DEQ) will be used in which participants rate acute responses to the e-cigarette on a 0-100mm scale from "not at all" (0mm) to "extremely" (100mm).
Irritation/Harshness: Score change in irritation of harshness of each e-cigarette condition (5 conditions in total) | Following administration of e-cigarette condition 1 (at 10 minutes), following administration of e-cigarette condition 2 (at 40 minutes)...following administration of e-cigarette condition 6 (at 160 minutes)
  Difference in irritation at each e-cigarette condition as measured by the computerized Generalized Labeled Magnitude Scale (gLMS). Participants will self-report their responses using a computer mouse to indicate where on the scale response falls. The Generalized Labeled Magnitude Scales (gLMS) are category ratio scales with seven semantic labels: "no sensation", "barely detectable", "weak", "moderate", "strong", "very strong", and "strongest imaginable", positioned quasi-logarithmically as per empirically determined semantic magnitudes on a 0-100 scale (strongest imaginable at the 100 end).

SECONDARY OUTCOMES:
Craving: Change in craving score for e-cigarette from baseline at each e-cigarette condition (5 conditions in total) | At baseline (at 0 minute), following administration of e-cigarette condition 1 (at 10 minutes), following administration of e-cigarette condition 2 (at 40 minutes)...following administration of e-cigarette condition 6 (at 160 minutes)
  Difference from baseline in craving for each e-cigarette condition will be measured by the Generalized Labeled Magnitude Scale (gLMS). Participants will self-report their craving for e cigarettes using a computer mouse to indicate where on the scale response falls. The Generalized Labeled Magnitude Scales (gLMS) are category ratio scales with seven semantic labels: "no sensation", "barely detectable", "weak", "moderate", "strong", "very strong", and "strongest imaginable", positioned quasi-logarithmically as per empirically determined semantic magnitudes on a 0-100 scale (strongest imaginable at the 100 end).
Changes of salivary Nicotine and Cotinine Levels from baseline at each e-cigarette condition (6 conditions in total) | At baseline (at 0 minute), Following administration of e-cigarette condition 1 (at 10 minutes), following administration of e-cigarette condition 2 (at 40 minutes)...following administration of e-cigarette condition 6 (at 160 minutes)
  Saliva samples will be collected following each exposure to product and before each lab sessions to assess change in nicotine/cotinine levels. These levels will be used for correlational analyses with behavioral measures and will be determined using LC/MS techniques at the core laboratory of university.

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, PhD, Principal Investigator — Yale University
Locations (1):
- JB Pierce Lab, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
We may share information about the IPD and study results with other researchers in the future, but the information will be de-identified.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The identifiable information will be kept for 7 years. After that, the data will become anonymous.
Access Criteria: The de-identified data will be made available for research purposes by contacting the PI.

REFERENCES:
- [Background] Lim J, Wood A, Green BG. Derivation and evaluation of a labeled hedonic scale. Chem Senses. 2009 Nov;34(9):739-51. doi: 10.1093/chemse/bjp054. PMID 19833660